CLINICAL TRIAL: NCT00198354
Title: Phase III Trial Comparing 2 Chemotherapy Schedules (Preoperative vs Pre and Postoperative) in Stage I and II NSCLC
Brief Title: Stage I/II NSCLC Perioperative Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-0002
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Non-small Cell Lung Cancer Stage I and II; Peri-operative Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A: pre-operative chemotherapy (Experimental): pre-operative chemotherapy (gemcitabine+cisplatine, 4 cycles)
  Interventions: Drug: gemcitabine + cisplatine
- B: pre-operative chemotherapy (Experimental): pre-operative chemotherapy (paclitaxel+carboplatin, 4 cycles)
  Interventions: Drug: gemcitabine + cisplatine
- C: peri-operative chemotherapy (Experimental): peri-operative chemotherapy (gemcitabine+cisplatine, 4 cycles)
  Interventions: Drug: Paclitaxel + Carboplatine
- D: peri-operative chemotherapy (Experimental): peri-operative chemotherapy (paclitaxel+carboplatin, 4 cycles)
  Interventions: Drug: Paclitaxel + Carboplatine

INTERVENTIONS:
Drug: gemcitabine + cisplatine — gemcitabine 1250 mg/m², D1+D8 cisplatine 80 mg/m², D1 (D1=D22)
  Arms: A: pre-operative chemotherapy; B: pre-operative chemotherapy
Drug: Paclitaxel + Carboplatine — paclitaxel 200 mg/m², D1 carboplatin AUC 6, D1 (D1=D22)
  Arms: C: peri-operative chemotherapy; D: peri-operative chemotherapy

SUMMARY:
The addition of chemotherapy to lung cancer surgery is now considered as the standard of care. Solid data support postoperative chemotherapy but only few results are available in the preoperative setting. To define which timing of perioperative chemotherapy offers the best survival improvement, the IFCT 0002 study is conducted in France.

DETAILED DESCRIPTION:
In this multicenter study, patients are randomized to receive either two preoperative chemotherapy cycles plus two additional preoperative cycles if they respond to chemotherapy, or two preoperative plus two postoperative cycles in case of response.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically NSCLC stade I or II Resectable disease WHO performance status of 2 or less

Exclusion Criteria:

NSCLC stage III or IV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2001-05; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Compare 3-Years survival | 3 years

SECONDARY OUTCOMES:
Compare Objective response rate | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alain Depierre, Pr, Principal Investigator — Intergroupe Francophone de Cancerologie Thoracique
Locations (1):
- CHU Besancon - Pneumologie, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Westeel V, Quoix E, Puyraveau M, Lavole A, Braun D, Laporte S, Bigay-Game L, Pujol JL, Ozenne G, Riviere A, Douillard JY, Lebeau B, Debieuvre D, Poudenx M, David P, Molinier O, Zalcman G, Lemarie E, Morin F, Depierre A, Milleron B; Intergroupe Francophone de Cancerologie Thoracique. A randomised trial comparing preoperative to perioperative chemotherapy in early-stage non-small-cell lung cancer (IFCT 0002 trial). Eur J Cancer. 2013 Aug;49(12):2654-64. doi: 10.1016/j.ejca.2013.04.013. Epub 2013 Jun 1. PMID 23735703
- [Result] de Fraipont F, Levallet G, Creveuil C, Bergot E, Beau-Faller M, Mounawar M, Richard N, Antoine M, Rouquette I, Favrot MC, Debieuvre D, Braun D, Westeel V, Quoix E, Brambilla E, Hainaut P, Moro-Sibilot D, Morin F, Milleron B, Zalcman G; Intergroupe Francophone de Cancerologie Thoracique. An apoptosis methylation prognostic signature for early lung cancer in the IFCT-0002 trial. Clin Cancer Res. 2012 May 15;18(10):2976-86. doi: 10.1158/1078-0432.CCR-11-2797. Epub 2012 Mar 20. PMID 22434665
- [Result] Mouillet G, Monnet E, Milleron B, Puyraveau M, Quoix E, David P, Ducolone A, Molinier O, Zalcman G, Depierre A, Westeel V; Intergroupe Francophone de Cancerologie Thoracique (IFCT). Pathologic complete response to preoperative chemotherapy predicts cure in early-stage non-small-cell lung cancer: combined analysis of two IFCT randomized trials. J Thorac Oncol. 2012 May;7(5):841-9. doi: 10.1097/JTO.0b013e31824c7d92. PMID 22722786
- [Result] Levallet G, Bergot E, Antoine M, Creveuil C, Santos AO, Beau-Faller M, de Fraipont F, Brambilla E, Levallet J, Morin F, Westeel V, Wislez M, Quoix E, Debieuvre D, Dubois F, Rouquette I, Pujol JL, Moro-Sibilot D, Camonis J, Zalcman G; Intergroupe Francophone de Cancerologie Thoracique (IFCT). High TUBB3 expression, an independent prognostic marker in patients with early non-small cell lung cancer treated by preoperative chemotherapy, is regulated by K-Ras signaling pathway. Mol Cancer Ther. 2012 May;11(5):1203-13. doi: 10.1158/1535-7163.MCT-11-0899. Epub 2012 Mar 12. PMID 22411898
- See also: Official website — http://www.ifct.fr